CLINICAL TRIAL: NCT07344285
Title: A Prospective Study of Cardiovascular Risk of Patients Admitted for Acute Exacerbation of COPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fanny W.S. Ko, Honorary clinical professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUHK_Resp_2026_Ko_01
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Patients with identified CV diseases will exhibit higher-risk profiles (e.g., elevated BMI, severe symptoms, frequent prior exacerbations), and the implementation of the care bundle will reduce re-admission rates compared to historical standard care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation of the COPD discharge care bundle (Experimental): Prospective recruitment with implementation of the COPD discharge care bundle
  Interventions: Procedure: Intervention Group
- Historic controls (Other): Historical records of prior acute exacerbation of COPD episodes and management under standard care from the database
  Interventions: Procedure: Usual Care

INTERVENTIONS:
Procedure: Intervention Group — Implementation of a COPD discharge care bundle for multidisciplinary support, providing optimal care for patients following acute exacerbations during hospital discharge.
  Arms: Implementation of the COPD discharge care bundle
Procedure: Usual Care — Patient undergoing usual care from historic controls
  Arms: Historic controls

SUMMARY:
This is a prospective study to assess the burden of existing or hidden cardiovascular (CV) and renal disease in patients with acute exacerbation of chronic obstructive pulmonary disease (AECOPD) in a Hong Kong public hospital setting. By implementing a chronic obstructive pulmonary disease (COPD) discharge care bundle with integrated CV/renal screening, the study aims to quantify undiscovered disease prevalence, evaluate risk factors for future exacerbations, and compare re-admission rates against historical controls, ultimately informing integrated cardiopulmonary management strategies.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a major global health concern, characterized by persistent respiratory symptoms and airflow limitation, and it frequently coexists with cardiovascular disease (CVD), which significantly contributes to morbidity and mortality in this population.

This is a prospective study to assess the burden of existing or hidden cardiovascular (CV) and renal disease in patients with acute exacerbation of COPD (AECOPD) in a Hong Kong public hospital setting. By implementing a COPD discharge care bundle with integrated CV/renal screening, the study aims to quantify undiscovered disease prevalence, evaluate risk factors for future exacerbations, and compare re-admission rates against historical controls, ultimately informing integrated cardiopulmonary management strategies.

The objectives and hypotheses are as follows:

Objectives and Hypotheses Primary Objective To describe the prevalence of undiscovered cardiovascular and renal disease burden among patients hospitalized for AECOPD in a Hong Kong public clinical setting.

• Hypothesis: A significant proportion of AECOPD patients will have previously undiagnosed CV or renal diseases identified through proactive screening, highlighting the need for routine assessments.

Secondary Objectives

1. To describe the pattern of AECOPD risk factors among COPD patients.
2. To describe the hospital re-admission rate after care optimization. • Hypotheses: Patients with identified CV diseases will exhibit higher-risk profiles (e.g., elevated BMI, severe symptoms, frequent prior exacerbations), and the implementation of the care bundle will reduce re-admission rates compared to historical standard care.

Exploratory Objectives

1. To describe the hospital re-admission rate after care optimization according to the cause of hospitalization (e.g., COPD exacerbation vs. CV/renal-related causes).
2. To describe the change in COPD treatment before and after care optimization. • Hypotheses: Re-admissions will be lower for CV/renal causes post-optimization, and a notable percentage of patients will require medication adjustments, such as escalation of inhaler or cardio-kidney-metabolic medications.

The COPD discharge care bundle includes:

1. COPD treatment optimization (per Global Obstructive Lung Disease [GOLD] 14 recommendations).
2. CV and renal disease check-up (NT-proBNP, Hba1c, troponin, eGFR, uACR, blood pressure and ECG).
3. Early follow-up at weeks 4-8.
4. Inhaler technique review and education. Patients with newly screened/diagnosed CV or renal diseases will be managed per routine clinical practice according to the relevant international guidelines, with referrals to cardiologists as needed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 years
* Patients hospitalized due to COPD exacerbation.
* Patients diagnosed with COPD, a confirmed COPD diagnosis with a specific FEV1/FVC ratio (<0.70)
* Able to provide informed consent

Exclusion Criteria:

* Pregnant subjects
* Inability to give informed consent
* Cancer patient who are on active chemotherapy or on palliative care

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2029-01-16 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients observed to have different high-risk factors for future COPD exacerbation | 12 months
  Percentage of patients observed to have different high-risk factors for future COPD exacerbation

SECONDARY OUTCOMES:
Re-admission rate | 12 months
  Re-admission rate due to COPD/cardiovascular/renal-related causes
Major Adverse Cardiac Events (MACE) | 12 months
  Major Adverse Cardiac Events (MACE), defined as myocardial infarction, stroke, death due to cardiovascular events, heart failure, arrhythmias, target vessel revascularization (e.g., repeat angioplasty), unscheduled coronary revascularization and cardiac arrest, will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: David SC Hui, MD, Study Director — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is available to qualified investigators upon reasonable request. Interested parties should submit a proposal outlining the intended use of the data. Requests will be evaluated for scientific merit and alignment with ethical guidelines. Approved data will be transferred through secure, encrypted channels under a formal data-sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From 17 Jan 2026 to 17 Jan 2046
Access Criteria: The principal investigator will access the IPD and supporting information.